CLINICAL TRIAL: NCT07145489
Title: An Open Label Pilot Study of Infrared Photobiomodulation in Humans With Epilepsy
Brief Title: Infrared Photobiomodulation in Humans With Epilepsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Goldenholz, Assistant Professor, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025P000606
Record Dates: First submitted 2025-08-19; First posted 2025-08-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Drug Resistant Epilepsy
Keywords: epilepsy; photobiomodulation; seizure
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsy; Seizures | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- photobiomodulation (Experimental): participants will use photobiomodulation daily for 6 months
  Interventions: Device: photobiomodulation

INTERVENTIONS:
Device: photobiomodulation — a hat with infrared lights will be worn for 30 minutes daily for 6 months

SUMMARY:
Drug-resistant epilepsy represents roughly 40% of people with epilepsy. It is very challenging to stop seizures in this condition, and the treatment options are limited. This study aims to investigate a new treatment that involves using infra-red light. In animals, this treatment has shown promise as a possible way to reduce seizures, but it has not been tested in humans for this. The investigators are interested to know if it can reduce seizures, and how comfortable it is to be treated with this therapy.

DETAILED DESCRIPTION:
Epilepsy affects 12 out of every 1000 people in the United States (1.2%). Of those, roughly 40% have drug-resistant epilepsy, meaning seizures do not stop despite good doses given with two different anti-seizure medications. Patients in this situation have several options (1) try additional medications (2) consider surgery to remove the part of the brain causing seizures, if possible (3) consider neuromodulation devices that change the brain activity using electricity in the brain (also a surgery) (4) try special diets such as the ketogenic diet which changes the fuel used by the brain by only eating certain foods. Despite these options, a large number of patients continue to have seizures. There is a great need for new treatments for drug resistant epilepsy.

The main purpose of this study is to determine if a new treatment is safe and well tolerated. Everyone in this study will receive the Red Light Therapy Hat which is investigational and is not approved by the FDA. The investigators do not know all the ways that this study treatment may affect people. This study is intended to hopefully help the participants, and the investigators hope the information from this study will help us develop a better treatment for drug resistant epilepsy in the future.

This particular investigational technology has been approved by the FDA for use in other diseases or conditions, but the investigators do not yet know if it is useful or safe as a treatment for drug resistant epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Drug resistant epilepsy
* Age 18 or older
* Average seizure rate of at least 2 seizures per month
* Accurate seizure diary with at least 3 months recorded

Exclusion Criteria:

* Implanted intracranial neurostimulation device (DBS or RNS)
* Intracranial shunt
* Skin photosensitivity
* Cancer on scalp
* Taking any medication that can cause photosensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2026-09-25 (Estimated); Study Completion 2027-09-25 (Estimated)

PRIMARY OUTCOMES:
seizure rate reduction | 6 months
  fraction of seizures reduced by therapy assessed by individual baseline rate
tolerability of daily photobiomodulation | 6 months
  Do participants find it reasonable to use the therapy daily or do they request exiting from the study? Do participants report significant side effects as reported by weekly check-ins that make the therapy uncomfortable or intolerable?

SECONDARY OUTCOMES:
seizure duration | 6 months
  fraction of seizure duration reduction assessed by baseline seizure durations

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Goldenholz, MD PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- BIDMC, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data about seizure rates, seizure durations and side effects
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: 1 year after the completion of enrollment, and for at least 4 years thereafter
Access Criteria: It will be made publicly accessible to anyone via public repository and via journal publication